CLINICAL TRIAL: NCT05836701
Title: Single-center Retrospective Study of Germ Cell Tumors of the Central Nervous System
Brief Title: Retrospective Study of Germ Cell Tumors of the Central Nervous System
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Junping Zhang, Director of Neuro-Oncology, Beijing Sanbo Brain Hospital
Other Study IDs: CNS-GCT-R
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Germ Cell Tumor of CNS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Retrospectively analyzing the epidemiological and clinical characteristics, treatment, recurrence, prognosis and prognostic factors of the germ-cell tumors of central nervous system in a single center.

DETAILED DESCRIPTION:
Clinical data of patients with germ-cell tumors of central nervous system who were treated in the Department of Neuro-oncology, Sanbo Brain Hospital Capital Medical University between January 2007 and December 2022 were retrospectively collected, and the epidemiological and clinical characteristics, treatment, recurrence, prognosis and prognostic factors of the disease were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Clinically or pathologically diagnosed as germ cell tumor of the central nervous system.
* Have received antitumor therapy.
* Patients who were clinically diagnosed based on neuroimaging characteristics and response to radiotherapy or chemotherapy were allowed for enrollment.

Exclusion Criteria:

* Patients with missing key information such as tumor location, surgical, chemotherapy and radiotherapy data, and post-treatment evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sanbo Brain Hospital, Capital Medical University
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
epidemiological characteristics | 1 year
treatment regimen | 1 year
relapse pattern | 1 year
prognostic factor | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jun-ping Zhang, Principal Investigator — Capital Medical University
Locations (1):
- Sanbo Brain Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No